CLINICAL TRIAL: NCT06395272
Title: Effects of Proprioceptive Sensitivity Stimulation Via the SURA Electrodevice on Kinematics, Kinetics and Spatiotemporal Parameters of Gait: a Pilot Study.
Brief Title: Effects of Proprioceptive Sensitivity Stimulation Via the SURA Electrodevice on Kinematics, Kinetics and Spatiotemporal Parameters of Gait.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-04-18
Record Dates: First submitted 2024-04-21; First posted 2024-05-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The design is a prospective longitudinal randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL (Experimental): The first phase of the intervention (device-on rest phases) will consist of the activation of the device on the muscle motor points of the medial belly of the gastrocnemius, soleus and peroneus muscles.The second phase (OFF activity-device phase) consists of carrying out the therapy as the patient had been doing normally in the Neurorehabilitation department at the center at a rate of 3 sessions per week on an outpatient basis according to their individualized needs.
  Interventions: Device: SURA
- COMPARATOR (Sham Comparator): The first phase of the intervention (device-on rest phases) will consist of the activation of the device on the muscle motor points of the medial belly of the gastrocnemius, soleus and peroneus muscles.The second phase (OFF activity-device phase) consists of carrying out the therapy as the patient had been doing normally in the Neurorehabilitation department at the center at a rate of 3 sessions per week on an outpatient basis according to their individualized needs.The control group will perform the same activity, but without the device activated during the device-on rest phases and adapted to the needs of each participant in their usual sessions without a standardized protocol.
  Interventions: Device: SURA

INTERVENTIONS:
Device: SURA — The motor points are the site of penetration of the motor nerve fibres and the highest concentration of motor plates in the muscle, which when stimulated produce the maximum effective muscle contraction. For 15 minutes and in a comfortable seated position at 90° hip, knee and foot, sustained pressure of 30 seconds each shall be exerted through the output plunger of the proprioceptive stimulus device.

SUMMARY:
Recovery of function in people with central nervous system (CNS) injury after stroke is very much like a relearning process that takes advantage of preserved sensorimotor circuits. Relearning can be optimised by providing appropriate proprioceptive (or deep sensory) information to the spinal cord with the aim of maximally engaging the preserved neural circuits. The development of the SURA electrodevice offers this sensitive input mechanism, within the Botton Up therapies. And through research on its use, the impact on the different dimensions related to gait and its components, and the translation to the functional reality of the person, will be evaluated.

DETAILED DESCRIPTION:
Objective: To assess whether the SURA electrodevice improves relevant aspects of dynamic balance in stroke survivors.

Methods:The design is a prospective longitudinal randomised controlled trial with simple masking by the examiner to be carried out at the facilities of the Ricard i Fortuny Social and Health Centre (CSSV RiF). The first phase of the intervention (device-on rest phases) will consist of the activation of the device on the muscle motor points of the medial belly of the gastrocnemius, soleus and peroneus muscles. The motor points are the site of penetration of the motor nerve fibers and the highest concentration of motor plates in the muscle, which when stimulated produce the maximum effective muscle contraction. The second phase (OFF activity-device phase) consists of carrying out the therapy as the patient had been doing normally in the Neurorehabilitation department at the center at a rate of 3 sessions per week on an outpatient basis according to their individualized needs.

The control group will perform the same activity, but without the device activated during the device-on rest phases and adapted to the needs of each participant in their usual sessions without a standardized protocol.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hemispheric stroke (ischaemic or haemorrhagic) diagnosed by MRI or CT scan, at least 3 months after onset of stroke
* Ability to walk at least 10m (irrespective of the need for assistance)
* Weakness in ankle dorsiflexion of the paretic limb (TFM>3)
* Ankle ROM >30° and 0° of foot dorsiflexion in knee extension
* Age between 18 and 85 years
* Mini-Mental State Examination (MMSE) > 24 score, non-disabling cognitive impairment
* Presence of clonus and hyperresistance to passive joint movement.

Exclusion Criteria:

* Diagnosis of Cognitive, visual or cardiorespiratory disorder (including cardiac pacemaker placement, heart failure and arrhythmia)
* Orthopaedic intervention for IE
* Balance disorders with vestibular features
* Skin diseases
* Botulinum toxin treatment within the last year.
* In addition, subjects who had participated in other studies in the last six months that could interact with the current study will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
The kinematics, kinetics and spatio-temporal parameters of gait. | Start of intervention, at 4 weeks and at completion 8 weeks
  An instrumented gait analysis will be performed to obtain a set of spatiotemporal, kinematic and kinetic measurements.The movement will be captured by the Ephion Vitality system. The system consists of two pressure templates and seven inertial sensors (measuring linear acceleration, angular velocity and magnetic field in all three dimensions).

SECONDARY OUTCOMES:
Neuromuscular Activation | Start of intervention, at 4 weeks and at completion 8 weeks
  Neuromuscular Activation Myontec surface electromyograph with sensors will collect the electrical activity of the lower limb muscles involved in gait coactivation. (Activation of motor units in milliseconds)

OTHER OUTCOMES:
Maximum isometric force | Start of intervention, at 4 weeks and at completion 8 weeks
  Maximum isometric force Measurement in Newtons of the muscle groups of hip extensors and flexors, hip internal and external rotators, hip abductors and adductors, knee flexors and extensors, dorsiflexors and plantar flexors of the foot, foot inverters and eversors with K-Force Muscle Controller Kinvent manual muscle dynamometry.

CONTACTS AND LOCATIONS:
Locations (1):
- CSSV-Rif, Barcelona, Vilafranca Del Penedés, Spain

IPD SHARING:
Plan to Share IPD: No